CLINICAL TRIAL: NCT04306991
Title: Modifications of Heart Murmurs and Cardiac Output During Fever
Acronym: FeMur
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC19_0202
Record Dates: First submitted 2020-01-17; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2019-12

CONDITIONS: Heart Murmurs; Fever
MeSH Terms: conditions — Heart Murmurs; Fever

STUDY DESIGN:
Intervention Model Description: Each patient will be auscultated twice:
  * during a febrile episode (body temperature >38.5°C)
  * after resolution of fever (body temperature < 37.5°C)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Fever (Experimental): Auscultation using an electronic stethoscope Measurement of cardiac output using echocardiography
  Interventions: Device: Auscultation using an electronic stethoscope (EKO CORE 4)
- Apyrexia (Experimental): Auscultation using an electronic stethoscope Measurement of cardiac output using echocardiography
  Interventions: Device: Auscultation using an electronic stethoscope (EKO CORE 4)

INTERVENTIONS:
Device: Auscultation using an electronic stethoscope (EKO CORE 4) — * Auscultation using an electronic stethoscope (EKO CORE 4). Record of at least 3 cardiac cycles.
  * Measurement of cardiac output using echocardiography.

SUMMARY:
The combination of fever and auscultation of a heart murmur suggests the diagnosis of endocarditis. However, fever itself increases cardiac output and could therefore modify heart sounds. The aim of the FeMur study is to measure the modification of heart sounds during fever.

Heart sounds of 15 hospitalized febrile patients with a heart murmur will be recorded using an electronic stethoscope before and after resolution of fever. The records will be analyzed using a computerized application in order to quantify the intensity of heart murmurs.

DETAILED DESCRIPTION:
Fever is an frequently observed during acute illnesses, particularly infectious diseases. The hemodynamic consequences of fever have been extensively studied. Fever leads to an acceleration of heart rate (approximately 8.5 bpm per degree celsius) and to a moderate drop in blood pressure. Cardiac output increases in the context of heat stress as a result of complex physiological adaptations, including heart rate and systolic function increase while preload and after load decrease.

However, there are no studies on the specific consequences of fever on heart sounds. The question is important since auscultation of a heart murmur in a febrile patient suggests the diagnosis of endocarditis. In endocarditis, the heart murmur, which is present in 85% of cases, is due to the mutilation of heart valves, which requires urgent diagnostic and therapeutic management. Suspicion of endocarditis requires emergency cardiac ultrasonography. However, the proportion of patients with actual endocarditis among patients with heart murmur and fever is low. This could arise from the fact that fever itself may increase or trigger a heart murmur. Indeed, any increase in cardiac output may generate audible turbulence when blood is pumped across a heart valve.

Functional or inorganic murmurs are murmurs triggered by changes in cardiac output or blood viscosity, as opposed to organic murmurs reflecting an anatomical abnormality in the heart. Certain characteristics of the murmur and the context of occurrence can guide the clinical toward one of these two situations, but distinguishing functional from organic murmurs is most often difficult.

The impact of fever on cardiac murmurs has not been experimentally demonstrated. This is the aim of the FeMur study.

For this purpose, heart sounds of 15 patients will be recorded during a febrile ilness and after resolution of fever using an electronic stethoscope and analyzed using a computer application. The average intensity of heart murmurs will be compared between the two periods in order to determine the impact of fever.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized febrile patients (body temperature > 38.5°C)
* Aged 18 or older
* Agreement to participate to the study

Exclusion Criteria:

* Patients treated with beta-blockers, verapamil, or diltiazem
* Patients with atrial fibrillation
* Pregnancy or breastfeeding
* Patients with severe psychiatric disorder
* Patients with diminished heart sounds

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Murmur intensity | up to 7 days
  Proportion of patients with a modification of heart sounds (computerized comparison of murmur intensity during fever and during apyrexia)

SECONDARY OUTCOMES:
Cardiac output (echocardiography) | up to 7 days
  Comparison of cardiac output measured using echocardiography during fever and after resolution of fever (apyrexia)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Dubee, MD, PhD, Study Director — University Hospital, Angers

IPD SHARING:
Plan to Share IPD: No